CLINICAL TRIAL: NCT04394845
Title: Assessment of the Biodistribution and Safety of [18F]GTP1 in Healthy Japanese Subjects
Brief Title: A Study of the Biodistribution and Safety of [18F]GTP1 in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Invicro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GN42043
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Results first posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]GTP1 (Experimental): Participants will receive a single bolus injection of radioligand [18F]GTP1 intravenously (IV).
  Interventions: Diagnostic Test: [18F]GTP1

INTERVENTIONS:
Diagnostic Test: [18F]GTP1 — [18F]GTP1 IV bolus injection of up to 370 megabecquerel (MBq) (10 millicurie [mCi]), with a maximum drug mass dose of 10 microgram (μg).
  Other Names: [18F]G02941054

SUMMARY:
The purpose of this study is to evaluate the biodistribution, safety and tolerability of a single dose of [18F]GTP1 as a tau targeted radiopharmaceutical in healthy Japanese participants.

ELIGIBILITY:
Key inclusion criteria:

* Healthy with no clinically relevant finding on physical examination at screening and prior to radiopharmaceutical administration
* Female participants must be willing to avoid pregnancy and refrain from donating eggs during the treatment period and for 30 days after the final dose
* Male participants with partners of childbearing potential must commit to the use of two methods of contraception for the study duration and 90 days after the last dose
* Male participants must not donate sperm for the duration of the study and 90 days after the last dose
* Participants must have both Japanese parents and all Japanese grandparents

Key exclusion criteria:

* Participants with any significant medical disorder or disease expected to interfere with the study
* Current or prior history (within a six-month period) of exposure to nicotine products
* History of drug or alcohol abuse within 12 months prior to screening
* Prior participation in other research protocols or clinical care in the last year, such that radiation exposure combined with that from the present study exceeds an effective dose of 50 millisievert (mSv), the allowable annual limit for research participants as established by the US Federal Guidelines
* Use of any prescription drugs, herbal supplements, within 4 weeks prior to initial dosing
* Use of over the counter (OTC) medication, dietary supplements, or vitamins, within 2 weeks prior to initial dosing
* Known hypersensitivity to any component of the formulation of [18F]GTP1 or related compounds
* Major surgery, or donation or loss of 400 mL or more of blood within 4 weeks prior to initial dosing
* History of immunodeficiency diseases, including positive human immunodeficiency virus (HIV) test
* Positive for Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody
* Women who are pregnant, lactating or breastfeeding
* Unsuitable veins for repeated venipuncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Invicro, a Konica Minolta company, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening assessments were completed within 30 days of Day 1.
Groups:
- [18F]GTP1: Participants received a single bolus injection of radioligand [18F]GTP1 intravenously (IV).
Period: Overall Study
Arm/Group | [18F]GTP1
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | [18F]GTP1
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.33 (15.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: Kg] | 55.32 (11.29)

OUTCOME MEASURES:

1. Primary Outcome: Total Source Organ Counts Based on Individualized Organ Volumes of Interest (VOIs)
Description: Decay corrected [18F]GTP1 time-activity in the source organs acquired following bolus tracer injection and expressed as %Injected Dose (ID).
Time Frame: Day 1
Population: One participant was excluded from the analysis at mean collect times: 16.38604 and 32.41194 minutes due to power surge during the scan that caused the system to power off. The process to restart took ~20 min and the absence of these specific data points. There was no impact on the quality of the subsequent data.
Measure: Mean (Standard Deviation); unit: Percentage of Injected Dose
Arm/Group | [18F]GTP1
Number analyzed (Participants) | 6
Percentage of Injected Dose
  Mean collect time: 5.32767 minutes | 0.33530 (0.18795)
  Mean collect time: 16.38604 minutes: number analyzed (Participants) | 5
  Mean collect time: 16.38604 minutes | 0.59398 (0.11540)
  Mean collect time: 32.41194 minutes: number analyzed (Participants) | 5
  Mean collect time: 32.41194 minutes | 2.13730 (0.76985)
  Mean collect time: 53.21428 minutes | 4.89330 (1.41690)
  Mean collect time: 78.27645 minutes | 9.38103 (3.07024)
  Mean collect time: 97.78638 minutes | 12.93725 (4.91340)
  Mean collect time: 144.06733 minutes | 20.76320 (5.05449)
  Mean collect time: 187.27612 minutes | 25.22968 (6.09050)
  Mean collect time: 213.49112 minutes | 29.06417 (9.29250)
  Mean collect time: 258.12780 minutes | 34.50070 (9.38550)
  Mean collect time: 304.21875 minutes | 36.95242 (10.99721)
  Mean collect time: 337.49112 minutes | 39.75663 (10.21783)

2. Primary Outcome: Source Organ Residence Time (Total Number of Disintegrations)
Description: Source organ uptake and washout with calculation of total number of disintegrations (or residence time, or kinetic values) using the area under the time-activity curve divided by the injected dose of radiopharmaceutical
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: MBq x hour/MBq
Groups:
- [18F]GTP1 Female; [18F]GTP1 Male: Participants received a single bolus injection of radioligand [18F]GTP1 intravenously (IV).
Arm/Group | [18F]GTP1 Female | [18F]GTP1 Male
Number analyzed (Participants) | 3 | 3
MBq x hour/MBq
  Brain | 0.0375 (0.00295) | 0.0315 (0.00717)
  Gallbladder Contents | 0.0254 (0.038) | 0.0304 (0.023)
  Gallbladder Contents with GB emptying model | 0.0102 (0.012) | 0.0122 (0.00637)
  LLI Cont. | 0.0416 (0.00214) | 0.0396 (0.00401)
  SI Cont. | 0.415 (0.0219) | 0.395 (0.0397)
  ULI Cont. | 0.228 (0.0117) | 0.217 (0.0219)
  Heart Wall | 0.0153 (0.00326) | 0.019 (0.00774)
  Kidneys | 0.046 (0.0195) | 0.0448 (0.0114)
  Liver | 0.591 (0.112) | 0.532 (0.0284)
  Lungs | 0.0346 (0.00205) | 0.0523 (0.0125)
  Spleen | 0.00634 (0.00203) | 0.0074 (0.00339)
  Urinary Bladder Contents | 0.135 (0.047) | 0.237 (0.0332)
  Urinary Bladder Contents with UB voiding model | 0.18 (0.0717) | 0.222 (0.0441)
  Remainder | 0.743 (0.143) | 0.687 (0.056)
  Remainder with UB voiding model | 0.708 (0.181) | 0.675 (0.127)
  Remainder with both UB voiding and GB emptying models | 0.723 (0.161) | 0.693 (0.12)

3. Primary Outcome: Mean Radiation Absorbed Dose Estimates in Target Organs and Whole Body Based on Standard Medical Internal Radiation Dose (MIRD) Methodology
Description: Radiation absorbed dose estimates based on the Medical Internal Radiation Dose (MIRD) methodology utilizing urine data and International Commission on Radiological Protection (ICRP) gastrointestinal (GI) tract kinetics
Time Frame: Day 1
Population: Testes not analyzed for female population.
Measure: Mean (Standard Deviation); unit: mSv/MBq
Arm/Group | [18F]GTP1 Female | [18F]GTP1 Male
Number analyzed (Participants) | 3 | 3
mSv/MBq
  Adrenals | 0.0164 (0.00156) | 0.0123 (0.000451)
  Brain | 0.00789 (0.00075) | 0.00606 (0.00132)
  Breasts | 0.00595 (0.000974) | 0.00457 (0.00044)
  Gallbladder Wall | 0.0756 (0.0662) | 0.0713 (0.0353)
  LLI Wall | 0.0447 (0.00236) | 0.0376 (0.00314)
  Small Intestine | 0.117 (0.00513) | 0.0925 (0.00864)
  Stomach Wall | 0.0141 (0.000929) | 0.0106 (0.000758)
  ULI Wall | 0.127 (0.00513) | 0.105 (0.00974)
  Heart Wall | 0.0196 (0.00309) | 0.0167 (0.00439)
  Kidneys | 0.0429 (0.0119) | 0.037 (0.00705)
  Liver | 0.101 (0.0183) | 0.0702 (0.0034)
  Lungs | 0.0145 (0.000833) | 0.0138 (0.00191)
  Muscle | 0.0093 (0.000663) | 0.00732 (0.000499)
  Ovaries | 0.0276 (0.00133) | 0.0216 (0.00379)
  Pancreas | 0.0167 (0.00150) | 0.0128 (0.000379)
  Red Marrow | 0.0104 (0.000636) | 0.00841 (0.000637)
  Osteogenic Cells | 0.0107 (0.00161) | 0.00787 (0.000946)
  Skin | 0.0055 (0.000749) | 0.00428 (0.000441)
  Spleen | 0.0156 (0.00253) | 0.0133 (0.00313)
  Testes: number analyzed (Participants) | 0 | 3
  Testes |  | 0.00606 (0.000261)
  Thymus | 0.00667 (0.00117) | 0.00513 (0.00064)
  Thyroid | 0.00472 (0.00107) | 0.00388 (0.00064)
  Urinary Bladder Wall | 0.129 (0.0472) | 0.112 (0.0198)
  Uterus | 0.0258 (0.00225) | 0.0213 (0.0007)
  Total Body | 0.0134 (0.000808) | 0.0103 (0.000552)
  Effective dose (ED, ICRP-60) | 0.0303 (0.0008) | 0.0245 (0.000436)

4. Primary Outcome: Percentage of Participants With Adverse Events
Description: An AE is the appearance or worsening of any undesirable sign, symptom, or medical condition, even if the event is not considered to be related to study drug. Study drug includes the investigational drug under evaluation during any phase of the study. Medical conditions/diseases present before starting study drug are only considered AEs if they worsen after starting study drug. Abnormal laboratory values or test results constitute AEs only if they induce clinical signs or symptoms, are considered clinically significant, or require therapy.
Time Frame: Up to 5 days
Measure: Number; unit: Participants
Arm/Group | [18F]GTP1
Number analyzed (Participants) | 6
Participants | 1

ADVERSE EVENTS:
Time Frame: Baseline up to 5 days
Arm/Group | [18F]GTP1
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [18F]GTP1 (N=6)
Haematoma (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT04394845/Prot_SAP_000.pdf